CLINICAL TRIAL: NCT01988480
Title: Clinical Assessment of Innovative Procedure Using Image-guided Surgery to Avoid Sinus Lift
Brief Title: Guided Surgery Versus Sinus Graft
Acronym: SINIMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008.514
Record Dates: First submitted 2013-09-18; First posted 2013-11-20 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2020-06

CONDITIONS: Edentulous
Keywords: Guided surgery; Sinus graft
MeSH Terms: conditions — Mouth, Edentulous | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Image-guided surgery (Experimental): Image-guided implant placement
  Interventions: Procedure: Image-guided surgery
- sinus graft (Sham Comparator): Sinus lift surgery : Patients receive sinus graft before implant placement
  Interventions: Procedure: Sinus lift surgery

INTERVENTIONS:
Procedure: Image-guided surgery — Placement on residual bone around the implant
  Arms: Image-guided surgery
Procedure: Sinus lift surgery — Allograft bone
  Arms: sinus graft

SUMMARY:
The objective of this study is to compare two surgical procedure to place implant in severely resorbed posterioir part of the maxilla.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and more
* sinus lift
* enough remaining bone for image guided implant placement

Exclusion Criteria:

* pregnancy
* chronic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07-08 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Treatment success | 2 years
  Treatment success is defined as followed : a "yes" must be obtain for the 4 following item.
  * Each implant are placed as planned (location and time) before surgery for each patient
  * Implant stability for each implant at follow-up stage
  * No radiolucent image around each implant
  * No pain no infection and paresthesia around each implant

SECONDARY OUTCOMES:
Accuracy of the image guided system used | During surgery
  Implant placed or not
Treatment success | 5 years
Replacement of missing teeth | 4 month after surgery
Angulation of implant | 4 month after surgery
Cost of treatment | 4 month after surgery
  Medical economic aspect
Patient pain | 1 week after implant placement procedure
  Pain is evaluated by the patient using both a analogic visual scale ranging from 0 to 10 and qualitative data (null, moderate, important, severe).
  Time of pain evaluation:
  Arm: graft procedure
  * Day of graft procedure
  * 1 week after graft procedure
  * Day of implant placement (6 months after graft)
  * 1 week after implant placement
  Arm: image-guided surgery
  * Day of implant placement
  * 1 week after implant placement
Patient satisfaction | 1 year after prosthesis loading
  Satisfaction is evaluated using qualitative data after surgery (how unconfortable was the surgery: very hard, hard, not hard, no opinion) and 1 year after prosthesis loading (treatment fulfill your expectation: no - not satisfied - satisfied - very satisfied.
  After surgery (graft procedure and implant placement, the following question is also asked to the patient : would you recommend the surgical procedure to a friend.
  Time of satisfaction evaluation:
  Arm : graft procedure
  * 1 week after graft surgery
  * 1 week after implant placement
  * 1 year after prosthesis loading
  Arm : image-guided surgery
  * 1 week after surgery (implant placement)
  * 1 year after prosthesis loading

CONTACTS AND LOCATIONS:
Overall Officials: Thomas FORTIN, Principal Investigator — Hospices Civils de Lyon - Service de Consultations et Traitements Dentaires
Locations (1):
- Hospices Civils de Lyon - Service de Consultations et Traitements Dentaires, Lyon, France

REFERENCES:
- [Result] Almahrous G, David-Tchouda S, Sissoko A, Rancon N, Bosson JL, Fortin T. Patient-Reported Outcome Measures (PROMs) for Two Implant Placement Techniques in Sinus Region (Bone Graft versus Computer-Aided Implant Surgery): A Randomized Prospective Trial. Int J Environ Res Public Health. 2020 Apr 25;17(9):2990. doi: 10.3390/ijerph17092990. PMID 32344891